CLINICAL TRIAL: NCT03237884
Title: Reality Map of Integrated Oncology and Palliative Care in Romanian and Swiss Cancer Centres
Brief Title: Romanian-Swiss Research Programme IZERZO
Acronym: IZERZO
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Florian Strasser, MD ABHPM, Principal Investigator, Cantonal Hospital of St. Gallen
Other Study IDs: EKSG 13/157; IZERZO_142226/1 (Other Grant/Funding Number: Swiss National Foundation)
Record Dates: First submitted 2014-06-25; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-07

CONDITIONS: Advanced Incurable Cancer
Keywords: Palliative Care; Oncology; advanced incurable cancer (any type); integration; development; palliative care interventions; process indicators; Romania
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Palliative Care procedures should be integrated early in the course of disease of patients with advanced incurable cancer. With this study, where the investigators follow adult patients with incurable cancer over 6 months or until death (whatever occurs earlier), the investigators aim to identify patients' needs for Palliative Care interventions (like support in illness understanding and decision making, symptom management, concrete end-of-life preparation, and others) and their remembered delivery by health care professionals. The investigators also collect data on patients care (use of chemotherapy, intensive care in the last month of life) and quality of death and dying (assessed by post-death-interviews with bereaved relatives). The aim is to have a "reality map" on current integration of oncology and palliative care and to test if appropriate Palliative Care interventions predict a better outcome.

DETAILED DESCRIPTION:
Background The integration of Palliative Care (PC) in routine oncological care remains challenging, particularly in resource-restricted, culturally diverse, and regulatory/legal disperse settings like Romania. The investigators aim to collect original data ("reality map") about the implementation of Key-Interventions Palliative-Cancer-Care (KI-PCC) and specific outcome quality indicators (QI). The investigators also hypothesize that both predefined cofactors and appropriately delivered KI-PCC will predict quality of care.

Aim The aim is to detect gaps in the care of advanced incurable cancer patients. Because in this setting there are no predefined structures, the investigators focus on interventions perceived by the patient.

Methods The investigators' target population are advanced incurable cancer patients in different care settings (oncology clinics, Palliative Care centers, and hospice, varying in size, location (rural, urban) and grade of specialization) representing the heterogeneity of care in Romania. The investigators characterize the population using demographic data (EAPC basic dataset amended by country specific data like family structures and income), and validated tools for patient needs (IPOS, EQ5D). Need for and perceived Key interventions of Palliative Cancer Care (KI-PCC), measured by nurse-patient-interaction, are assessed. These KI-PCC include illness understanding, symptom management, decision making, spirituality, end-of-life-preparation, and network/family support. Further, the investigators collect defined outcome quality indicators (QI) for the integration (quality of death and dying, symptoms, aggressive end-of-life-care, inappropriate anticancer care, ER-visits). In addition, known, associated cofactors (e.g. comorbidities, living situation) are measured. The data collection will be longitudinal with monthly follow-ups for at most six months or until death. Focus groups at each participating center explore local influencing factors both for KI-PCC and QI. Several steps of quality assurance (source data verification, expert reviews of anticancer treatment, etc.) are introduced.

The analysis has three elements. First, the investigators will describe the population. Second, the investigators will map the patient perceived KI-PCC and defined outcome QI. Third, if data show robust after international expert review, the investigators will test the hypothesis that appropriate KI-PCC predict quality of care, measured by QI.

Expected impact The investigators expect that their approach will identify gaps in the integration of oncology and palliative care in their specific settings, focusing, however, mainly on patient and proxy view and backed by available information from outcome QI. The conduct of this protocol might also directly have an influence on patient care.

This approach will allow the development of tailored interventions in a next step. The investigators' approach may also serve as a model to measure the integration of oncology and palliative care in various settings, focusing on interventions.

ELIGIBILITY:
Inclusion Criteria:

* stage IV cancer
* over 18 years
* minimal symptom burden in IPOS (at least 3 symptoms over or equal 2)
* Eastern Cooperative Oncology Group (ECOG) Performance Status 1, 2, 3

Exclusion Criteria:

* cognitively impaired
* prognosis less than 1 month according to clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced, incurable cancer patients, adult, without cognitive impairment, with a minimal symptom burden (defined threshold on IPOS)
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Composite Endpoint | up to 6 months (or death, whichever occurs first)
  A composite endpoint, composed by the outcome indicators inappropriate anticancer care, repeated ER-admissions, high symptom burden (on IPOS), "aggressive" end-of-life-care, and bad quality of death and dying (QODD)

CONTACTS AND LOCATIONS:
Overall Officials: Florian Strasser, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (2):
- Oncological Institute "Prof. Dr. Ion Chiricuţă", Cluj-Napoca, Romania
- Kantonsspital St.Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided